CLINICAL TRIAL: NCT06516276
Title: Application of New Technologies to Improve the Quality of Life of Prostate Cancer Patients:
Brief Title: Technologies to Improve QoL of Prostate Cancer
Acronym: MIO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Inés Nuño de la Rosa García, Dr, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/38PI
Record Dates: First submitted 2024-07-12; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOBILE App (Experimental): The intervention group will receive standard nutrition, physical exercise, and emotional care recommendations according to scientific evidence and instructions on using the MIO mobile application.
  Interventions: Device: Mobile App M.I.O
- Control Standard Recommendations (No Intervention): The control group will receive the same recommendations without additional support tools.

INTERVENTIONS:
Device: Mobile App M.I.O — This mobile app provides patients with access to various resources and therapies focused on nutrition, exercise, and emotional well-being. The main objective is to measure the quality of life of the app users through validated questionnaires in a randomized health education study to evaluate whether a substantial improvement in their well-being is achieved.
  Arms: MOBILE App

SUMMARY:
The M.I.O Project, which stands for Comprehensive Oncological Medicine, aims to comprehensively and multidisciplinary address the effects of prostate cancer, specifically in patients with hormone-sensitive metastatic prostate cancer (HSMPC), an advanced stage of the disease that still offers prolonged survival due to new medications. The proposal seeks to develop a healthcare approach that promotes self-care and improves the physical and mental health of patients.

Despite growing scientific evidence supporting an integrative approach in oncological care, the provision of personalized options for exercise, nutrition, and psychological therapy before, during, and after diagnosis remains limited. The project proposes to develop tools such as a dedicated mobile application that provides HSMPC patients access to various resources and therapies to improve their health, focusing on nutrition, exercise, and emotional well-being.

M.I.O represents an innovative and holistic approach to addressing these patients' needs and improving their overall well-being. The main goal is to measure the quality of life of the application users through validated questionnaires in a randomized health education study to assess if there is a substantial improvement in their well-being.

ELIGIBILITY:
Inclusion Criteria:

* Patients histologically diagnosed with prostate cancer
* Metastases confirmed by validated imaging studies
* Not meet criteria for castration resistance.

Exclusion Criteria:

* Do not have a smartphone device
* Refuse to participate
* Not sign the informed consent.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure the quality of life of patients with metastatic prostate cancer using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). | At 3 and 6 months after use of the standard recommendatiosn/ Mobile App
  "Quality of life of patients with hormone-sensitive metastatic prostate cancer" refers to the well-being and daily functioning of individuals diagnosed with this condition, including their physical, emotional, and social health, and their ability to perform everyday activities despite cancer progression.
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) is a standardized tool used to assess cancer patients' quality of life. It includes 30 items covering physical functioning, emotional well-being, cognitive functioning, social interactions, and symptoms like fatigue and pain.
  Scores range from 0 to 100. Higher scores in functional scales and global health status indicate better functioning and quality of life, while higher scores in symptom scales/items indicate worse symptoms or problems.

SECONDARY OUTCOMES:
assess treatment adherence using the Morisky Medication Adherence Scale (MMAS) | At 3 and 6 months after use of the standard recommendatiosn/ Mobile App
  "Improving adherence to treatments" refers to enhancing patients' consistency in following prescribed medical regimens, such as taking medications correctly, attending scheduled appointments, and adhering to recommended lifestyle changes. The goal is to ensure that patients receive the full benefit of their treatments, leading to better health outcomes and more effective disease management. The Morisky Medication Adherence Scale (MMAS) is a validated questionnaire used to measure a patient's adherence to their medication regimen. It consists of a series of questions designed to identify patterns of behavior related to medication-taking.
  Scores range from 0 to 8. Higher scores indicate better adherence to the prescribed medication regimen. Specifically, for MMAS-8:
  A score of 8 suggests high adherence. A score of 6 to <8 indicates medium adherence. A score of <6 suggests low adherence.
Clinical progression using the Functional Assessment of Cancer Therapy - Fatigue (FACT-F) questionnaire and the Visual Analogue Scale (VAS). | At 3 and 6 months after use of the standard recommendatiosn/ Mobile App
  Assessing the impact of the application on clinical progression through pain and fatigue. The Functional Assessment of Cancer Therapy - Fatigue (FACT-F) questionnaire measures fatigue and its impact on quality of life in cancer patients, with scores ranging from 0 to 52; higher scores indicate better quality of life and less fatigue.
  The Visual Analogue Scale (VAS) measures subjective symptoms like pain or fatigue. It consists of a 10 cm line with "no pain" at one end and "worst pain imaginable" at the other. Patients mark their current state on the line, resulting in a score from 0 to 100; higher scores indicate greater symptom severity
Assessment of Compliance with Recommendations (Percentage Based on M.I.O. Application and Clinical Interview for Control Group) | At 3 and 6 months after use of the standard recommendatiosn/ Mobile App
  The objective is to measure the percentage of recommendations that were followed. This will be assessed using the M.I.O. application for the intervention group and through clinical interviews for the control group. The compliance rate will be calculated as the percentage of the total recommendations that each participant adhered to during the study period.

IPD SHARING:
Plan to Share IPD: Undecided